CLINICAL TRIAL: NCT05087017
Title: Influence of Regular Physical Activity on Sleep and Anxiety in Patients With Chronic Obstructive Pulmonary Disease and Idiopathic Lung Fibrosis
Brief Title: Influence of Regular Physical Activity on Sleep in Patients With COPD and Idiopathic Lung Fibrosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Other Study IDs: ACT.PHYS-001
Record Dates: First submitted 2021-09-08; First posted 2021-10-21 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Fibrosis, Pulmonary
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intervention Group: Patients with COPD or Lung Fibrosis following rehabilitation program will be invited to participate and answer the questionnaires in the beginning and after eight weeks of rehabilitation.
  Interventions: Other: Intervention group
- Control group: Patients with COPD or Lung Fibrosis who do not do any regular activity will be invited to participated and answer the questionnaires just once.

INTERVENTIONS:
Other: Intervention group — Patients with medical condition to follow the rehabilitation program will be asked to answer questionnaires to assess their sleep quality.
  Groups: Intervention Group

SUMMARY:
The study looked at whether regular physical activity can influence sleep duration, sleep quality and/or anxiety in patients with chronic obstructive pulmonary disease (COPD) and idiopathic pulmonary fibrosis (IPF).

The link between exercise and sleep has already been observed in the literature, but the impact of exercise on sleep is poorly understood. The question is how important is the influence of regular physical activity on sleep, anxiety and depression in patients with COPD or IPF.

DETAILED DESCRIPTION:
Patients will be selected in two ways:

1. Intervention group: patients with COPD or idiopathic fibrosis following rehabilitation program in our center, who meet the inclusion criteria will be invited to participate in the survey and answer the questionnaires during the first week and again eight weeks after the start of the rehabilitation program.
2. Control group: patients with COPD or idiopathic fibrosis who do not perform any regular physical activity will be invited to participate in the survey and answer the questionnaires.

The questionnaires are validated and the time allowed for completion is 45 minutes. The questionnaires will assess sleep quality, anxiety and symptoms of depression.

ELIGIBILITY:
Inclusion Criteria:

* Patients with COPD.
* Patients with Idiopathic Pulmonary Fibrosis.
* Patients who can read and write in French.
* Patients who agree to participate in research and sign the informed consent form.
* Patients who participated of our rehabilitation program or Patients who do not do any regular exercise activity.

Exclusion Criteria:

* Regular use of Continuous Positive Airway Pressure devices (CPAP)

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with COPD or lung fibrosis.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-02-20 (Actual); Primary Completion 2021-11-20 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
Changes in sleep quality - sleepiness | 2 minutes
  Sleep quality will be assessed by the questionnaire "Epworth Sleepiness Scale". A score between 0-5 indicates "lower normal daytime sleeping"; between 6-10 "higher normal daytime sleepiness; 11-12 "mil excessive daytime sleepiness"; 13-15 "moderate excessive daytime sleepiness" and 16-24 "severe excessive daytime sleepiness".
Changes in sleep quality - insomnia | 2 minutes
  Sleep quality will be assessed by the questionnaire "Insomnia Severity Index ". A scale is used to rank each item, where "0" means "no problem", "1 - mild problem", "2 - moderate" "3 - severe" and "4 very severe problem". The total score is interpreted as absence of insomnia (0-7); sub-threshold insomnia (8-14); Moderate insomnia (15-21); and severe insomnia (22-28).
Changes in sleep quality - "Morningness" or "eveningness" types | 2 minutes
  Sleep quality will be assessed by the questionnaire "Morningness - Eveningness Questionnaire ". Scores between 42 and 58 indicate "neural types", scores of 59 and above indicate "morning types" and scores of 41 and below indicates "evening types".
Changes in sleep quality - Sleep Agenda | 4 minutes per day
  Sleep quality will be assessed by the questionnaire "Sleep Agenda". The sleep agenda is a subjective method of sleep evaluation which demand the patient to fill the agenda at two times of the day: at 9 in the morning to describe what happened at night and 9 in the evening to report what happened in the day for a minimum of three weeks. The patient need to specify the quality of his night, if it was "very good", "good", "average", "bad" and "very bad" and specify, also, if he took any medications or if something happened may have interfered with his sleep.

SECONDARY OUTCOMES:
Changes in anxiety symptoms | 3 minutes
  Nijmegen Questionnaire is a valid questionnaire to detect patients who have hyperventilation symptoms which the complaints may not be fully due to physiological abnormality, that is, it reflects a subjective aspect of dysfunctional breathing reflecting anxiety symptoms. Scores > 23 is indicative of dysfunctional breathing.
Changes in back pain symptoms | 2 minutes
  Back pain will be assessed by the "STarT Back Screening Tool". It is a quick-to-use self-administered questionnaire (9 items) that classifies patients with low, medium or high risk of low back pain.
  The score higher than 5 represents high risk of low back pain.
Changes in back pain symptoms and disability | 2 minutes
  Back pain will be assessed by "Oswestry Disability Index". It gives a subjective percentage score of level of function (disability) in activities of daily living in those rehabilitating from low back pain.
  The score goes to 0 to 100 describing the level of disability. The higher the score, the greater the severity of disability.
Changes in depression symptoms | 2 minutes
  Depression symptoms will be assessed by "Beck Depression Inventory ". It is composed of 21 items of symptoms and attitudes depressives, each category describes a specific behavioral manifestation of depression.
  The score goes from 1 to 40 describing the level of depression. The higher the score, the greater the severity of depression.

CONTACTS AND LOCATIONS:
Locations (1):
- Cliniques universitaires Saint-Luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No